CLINICAL TRIAL: NCT07278388
Title: Motivated Decision-Making and Performance
Brief Title: Neural Mechanisms of Fatigue in Post-Acute Sequela of SARS-CoV-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00283000_1; R01NS140610 (NIH)
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: PASC Post Acute Sequelae of COVID 19; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PASC Participants - Physical Fatigue Task (Experimental): Participants will perform a physically demanding task (grip force exertion task) repeatedly to induce physical fatigue.
  Interventions: Behavioral: Physical Fatigue
- Control Participants - Physical Fatigue Task (Experimental): Participants will perform a physically demanding task (grip force exertion task) repeatedly to induce physical fatigue.
  Interventions: Behavioral: Physical Fatigue

INTERVENTIONS:
Behavioral: Physical Fatigue — Participants will perform a physically demanding task (grip force exertion task) repeatedly to induce physical fatigue.

SUMMARY:
This proposal aims to understand the neurobiological mechanisms of fatigue in individuals with Post-Acute Sequelae of SARS-CoV-2 Infection (PASC). This knowledge will eventually provide candidate mechanisms to target with pharmacological intervention and inform rehabilitative care for those individuals suffering from symptoms of fatigue in PASC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old.
* Have received a clinical diagnosis of post-acute sequelae of SARS-CoV-2 (PASC)/long COVID syndrome using the criteria specified by Thaweethai, et al., 2023 (JAMA). This symptom checklist provides a score based on the number and severity of symptoms. An individual with a score >12 is classified as having PASC.
* Currently experiencing Fatigue/Brain Fog as assessed with the Post-COVID symptom checklist and the PedsQL questionnaire.

Exclusion Criteria:

* Neurological disorders including, but not limited to, stroke, head injury, epilepsy, seizures, brain tumors, brain surgery, Parkinson's Disease, or any other neuromuscular disease (self-report).
* Diagnosed history of severe psychiatric diseases such as depression and schizophrenia (self-report).
* Congestive heart failure.
* Peripheral artery disease with claudication.
* Cancer.
* Pulmonary or renal failure.
* Unstable angina.
* Uncontrolled hypertension (more than 190/110 mmHg).
* Severe aphasia.
* Orthopedic or pain conditions.
* Have had exposure to metal or metal implants, due to the hazardous effects of the magnetic field.
* If on immunomodulatory therapy, they must have been on that therapy for at least 6 months before the start of the study.

Healthy age- and sex-matched controls for PASC - Exclusion criteria: Participants with a history of any of the following will be excluded from the study:

* Hospitalization due to SARS-CoV-2 infection.
* Neurological disorders including, but not limited to, stroke, head injury, epilepsy, seizures, brain tumors, brain surgery, Parkinson's Disease, or any other neuromuscular disease (self-report).
* Diagnosed history of severe psychiatric diseases such as depression and schizophrenia (self-report).
* Congestive heart failure.
* Peripheral artery disease with claudication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between PASC and HC - difference in mean Assessment Error | Baseline, during experimental protocol.
  The difference between the level of effort rated by participants, and their average grip force exerted on a grip force dynamometer. Compared between PASC and HC.
Comparing between PASC and HC - difference in BBB permeability | Baseline, during MRI acquisition.
  Collected from and MRI sequence designed to measure BBB permeability.
Comparing between PASC and HC - Regions of the brain that are sensitive to Assessment error as a function of disease state | Baseline, during experimental protocol.
  We will examine an fMRI contrast, at the time of effort assessment, between HC and PASC groups. This contrast will examine percent signal change in brain activity.
The modulatory effect of BBB permeability on the relationship between Neural Activity and Effort Assessment | Baseline, during experimental protocol and MRI aquisition.
  We will create a structural equation model that includes BBB permeability, fMRI activity, effort assessment behavior, and disease state (PASC/HC).
Comparing between PASC and HC - Difference in momentary subjective fatigue ratings | Baseline and during fatiguing exertions in the experimental protocol.
  Measures of subjective fatigue will be collected on self report scale that ranges from 'not fatigued at all' to 'very fatigued'.
Comparing between PASC and HC - Difference in Mean Acceptance Rate of Risky Effort Options between rested/baseline and fatigue choices | Baseline and during fatiguing exertions in the experimental protocol.
  Proportion of decisions in which inviduals choice to accept a risky effort opitions over a sure effort option.
Comparing between PASC and HC - Regions of the brain encoding a difference in effort cost between rested/baseline and fatigue choices | Baseline and during fatiguing exertions in the experimental protocol.
  We will examine a contrast between chosen effort value pre versus post fatigue, between the HC and PASC groups. This contrast will examine percent signal change in brain activity.
The modulatory effect of BBB permeability on the relationship between Neural Activity and change effort-based decision-making | Baseline, fatigueing exertion, and during experimental protocol and MRI aquisition
  We will create a structural equation model that includes BBB permeability, fMRI activity, change in effort-based decision-making, and disease state (PASC/HC).
Comparing between PASC and HC - Difference in mean assessment error as a function of time | Data collections at months 0, 3, 6, 12
  The difference between the level of effort rated by participants, and their average grip force exerted on a grip force dynamometer. Compared between PASC and HC.
Comparing between PASC and HC - Difference in momentary subjective fatigue ratings as a function of time | Data collections at months 0, 3, 6, 12
  Measures of subjective fatigue will be collected on self report scale that ranges from 'not fatigued at all' to 'very fatigued'.
Comparing between PASC and HC - difference in BBB permeability as a function of time | Data collections at months 0, 3, 6, 12
  Collected from and MRI sequence designed to measure BBB permeability.
Comparing between PASC and HC - Regions of the brain that are sensitive to Assessment error as a function of disease state and time | Data collections at months 0, 3, 6, 12
  We will examine a contrast, at the time of effort assessment, between HC and PASC groups, and use time as a covariate. This contrast will examine percent signal change in brain activity.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Chib, PhD, Principal Investigator — Johns Hopkins University; Kennedy Krieger Institute
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided